## Chronic coronary syndrome in Swedish primary care (COSPRI)

A cluster-randomized study on a single-visit package investigation versus routine sequential investigation for chronic coronary artery disease conducted in Swedish primary health care.

NCT ID:2022-04416-01

## Document revision history

| Issue | Summary of change |
|-------|-------------------|
| 01 | New document |

## Statistical considerations

Analyzes will be done according to the intention-to-treat principle.

Conventional descriptive methods of means (with standard deviations) or medians (with interquartile ranges) for continuous data and proportions for categorical data will be used to compile data.

Comparison between groups will be made using Chi-2 test for proportions and T-test or Mann

Whitney U test for continuous data, the latter if data are not normally distributed. The appropriate type of regression model will be used to estimate the relationship between waiting time and investigation model, package investigation or standard investigation. Due to cluster randomization mixed models will be used.

Downstream cardiac investigations, final outcome and cost per patient will be structured according to Table 1-3.

Table 1 Downstream cardiac investigations

| Modality | Package | standard |
|---|---|---|
| | investigation <sup>1</sup> | investigation <sup>2</sup> |
| | n= | n= |
| Myocardial | 0 | |
| perfusion scan, n (%) | | |
| perrusion scarr, ir (70) | | |

| Echocardiography | 0 | 0 |
|---------------------------------|---|---|
| Computed tomography angiography | | |
| Stress echocardiography | | |
| Magnetic resonance imaging | | |
| Invasive coronary angiography | | |
| Ergospirometry | | |
| ?? | | |

<sup>&</sup>lt;sup>1</sup> Myocardial perfusion scan, echocardiography and CT of heart.

Table 2 Final outcome after cardiac investigations

| Modality | Package | standard |
|----------------------|---------------|---------------|
| | investigation | investigation |
| | n | n |
| CORAI: | | |
| Significant coronary | | |
| artery stenosis. | | |
| CABG | | |
| PCI | | |
| Myocardial ischemia | | |
| Heart failure | | |
| EF < 50 % | | |
| Criteria for HFpEF: | | |
| EF>50 %, E/e'>15, | | |
| LAVI index >37 | | |
| mL/m <sup>2</sup> | | |
| Valve disease: | | |
| Aortic stenosis, > | | |
| 3m/sec | | |

<sup>&</sup>lt;sup>2</sup> Exercise stress bicycle test and echocardiography.

| Mitral insufficiency<br>with enlarged<br>cardiac chambers |
|-----------------------------------------------------------|
| Pulmonary<br>hypertension, > 3.2<br>m/sec |
| Dilated ascending aorta >45 mm |
| No signs of CAD |

Table 3

Cost per patient in total, per action, diagnosis or ruling out of CAD.

| Modality | Package | standard |
|---------------------|---------------|---------------|
| | investigation | investigation |
| | n | n |
| | n | n |
| All participants | | |
| CABG | | |
| PCI | | |
| Myocardial ischemia | | |
| Heart failure | | |
| Valve disease | | |
| No signs of CAD | | |